CLINICAL TRIAL: NCT03870828
Title: Incidence, Clinical Characteristics and Evaluation of Prognostic and Diagnostic Markers of Interstitial Pneumonia With Autoimmune Features (IPAF) - a Multicenter Prospective Study
Brief Title: Clinical Characteristics of Interstitial Pneumonia With Autoimmune Features (IPAF) - a Multicenter Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Adam Barczyk, Professor, Ph.D., M.D., Medical University of Silesia
Other Study IDs: SilesianMU1
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Interstitial Lung Disease; Interstitial Pneumonia; Interstitial Fibrosis; Autoimmune Diseases
Keywords: IPAF; CTD-ILD; ILD; diagnostic markers; progression markers
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis; Autoimmune Diseases | interventions — Walk Test; Blood Gas Analysis; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following biospecimens will be collected:
  * blood (whole venous blood and serum)
  * bronchoalveolar lavage fluid
  * samples of bronchial mucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group IPAF: Patients with IPAF which is defined according to the Work Group of the European Respiratory Society/American Thoracic Society.
  The interventions to be administered include:bronchoalveolar lavage and taking bronchial mucosa samples lung function tests,6 minute walk test, use of cough and dyspnea scales, transthoracic echocardiography, blood testing, arterial blood gas and pulse oximetry
  Interventions: Diagnostic Test: Bronchoalveolar lavage and taking bronchial mucosa samples; Diagnostic Test: 6minute walk test; Diagnostic Test: Arterial blood gas; Procedure: Blood drawing
- Control group CTD-ILD: Patients with connective tissue disease associated intestitial lung disease: rheumatoid arthritis - RA, systemic sclerosis - SSc, polymyositis - PM, dermatomyositis - DM, (anti-synthetase syndrome - AS, Sjögren's syndrome - SjS, mixed connective tissue disease - MCTD ,systemic lupus erythematosus - SLE, diagnosed according to diagnostic criteria issued by European League Against Rheumatism (EULAR) and/or American College of Rheumatology (ACR)
  Interventions: Diagnostic Test: Bronchoalveolar lavage and taking bronchial mucosa samples; Diagnostic Test: 6minute walk test; Diagnostic Test: Arterial blood gas; Procedure: Blood drawing
- Control group ILD: Idiopathic interstitial pneumonia group: idiopathic pulmonary fibrosis - IPF, nonspecific interstitial pneumonia - NSIP, cryptogenic organizing pneumonia - COP, acute interstitial pneumonia - AIP; respiratory bronchiolitis associated interstitial lung disease - RB-ILD, desquamative interstitial pneumonia - DIP, lymphocytic interstitial pneumonia - LIP).
  Interventions: Diagnostic Test: Bronchoalveolar lavage and taking bronchial mucosa samples; Diagnostic Test: 6minute walk test; Diagnostic Test: Arterial blood gas; Procedure: Blood drawing

INTERVENTIONS:
Diagnostic Test: Bronchoalveolar lavage and taking bronchial mucosa samples — Regional anesthesia and sedation with use of lidocaine and midazolam will be performed, according to anesthesia protocols applied in respective endoscopy units. Intravenous cannula will be inserted prior to BF. During endoscopy, the patient will be monitored according to safety protocols applied in respective endoscopy units.
  Bronchoalveolar lavage will be performed in the bronchus from the middle robe of right lung or the lingula of left lung (B4, B5). Localization will be chosen based on HRCT results and will be recorded in patient's medical history. Sterile solution of 0, 9% NaCl will be instilled. 200 ml fluid will be applied with a syringe in portions of 25 ml or 50 ml. It is recommended that minimum 60 % of the lavage fluid is retrieved.
Diagnostic Test: 6minute walk test — a submaximal exercise test which entails measurement of distance walked over a span of 6 minutes. Blood pressure, pulse oximetry are measured directly before and after the test. The participant is also periodically asked about their dyspnea sensation
  Other Names: 6MWT
Diagnostic Test: Arterial blood gas — If SpO2 is measured to be < 92%, an artery (radial or femoral) is punctured in order to take a sample of arterial blood. Then, the artery is compressed in order to prevent bleeding/ hematoma.
  Other Names: ABG
Procedure: Blood drawing — A vein will be punctured in order to take a blood sample for further tests

SUMMARY:
Interstitial pneumonia with autoimmune features (IPAF) was defined in 2015 by the Working Group of the European Respiratory Society (ERS) and the American Thoracic Society (ATS) as interstitial pneumonia with some clinical and/or serological features suggesting presence of an underlying autoimmune disorder. However, ofiicial criteria for diagnosis of an autoimmune disease are not met.

Aims of the study:

1. Determine the incindence of IPAF in comparison with interstitial lung diseases (ILDs) and classic autoimmune diseases (ADs) in polish pulmonological centers.
2. Clinical, serological, functional and radiological and histopathological characteristics of IPAF patients.
3. Analysis of diagnostic strategies towards specific IPAF subgroups.
4. Characterictics of potencial diagnostic, predictive and prognostic features of IPAF.
5. Prospective assessment of IPAF patients in the courseof 5 years in order to determine stability of the diagnosis and potential progression to other diseases, e.g. ADs.

DETAILED DESCRIPTION:
The following patient groups will be studied:

1. Study group - IPAF.
2. Control groups:

   1. Connective tissue disease associated interstitial lung disease (CTD-ILD) patients: .rheumatoid arthritis - RA, systemic sclerosis - SSc, polymyositis - PM, dermatomyositis - DM, (anti-synthetase syndrome - AS, Sjoegren's syndrome - SjS, mixed connective tissue disease - MCTD ,systemic lupus erythematosus - SLE, diagnosed according to diagnostic criteria issued by European League Against Rheumatism (EULAR) and/or American College of Rheumatology (ACR)
   2. Idiopathic interstitial pneumonia group: idiopathic pulmonary fibrosis - IPF, nonspecific interstitial pneumonia - NSIP, cryptogenic organizing pneumonia - COP, acute interstitial pneumonia - AIP; respiratory bronchiolitis associated interstitial lung disease - RB-ILD, desquamative interstitial pneumonia - DIP, lymphocytic interstitial pneumonia - LIP).

      Methods Patients will be assessed by a pulmonologist and rheumatologist. Questionnaires regarding clinical symptoms, concomitant diseases and their treatment, disease activity will be fulfilled.

      The majority of diagnostic tests and procedures are routinely performed during clinical care.

      The study will be divided into 2 phases:
      1. Phase 1 - visit 1
      2. Phase 2 - observation of selected subjects from visit 1 to 5

      Phase 1:

      30 patients meeting the eligibility criteria, including individuals with a long medical history and currently undergoing treatment for interstitial lung disease/ autoimmune disorder are going to be recruited to the study in every clinical center, totaling up to:
      * 210 patients in IPAF group
      * 210 patients in CTD-ILD group
      * 210 patients in IIP group

      Phase 2 Only newly diagnosed patients (individuals who have not been previously diagnosed with interstitial lung disease, and such diagnosis was set during phase 1 of the study) will be recruited to this phase. Due to rare incidence, the recruitment phase may take up to 36 months.

      The total number of patients will be
      * 70 in IPAF group
      * 70 in CTD-ILD group (RA, SSc, PM, DM)
      * 70 in IIP group (35 with IPF and 35 with NSIP, COP and LIP)

      Visit 1:

      • The following tests and procedures will be performed:
      * Detailed anamnesis obtained through 'visit 1 questionnaire' [non-routine procedure]
      * Lung function tests (spirometry with reversibility testing, plethysmography, diffusion lung capacity for carbon monoxide) [routine procedure]. Absolute value and % of the reference value will be assessed.

      FEV1 - Forced expiratory volume in 1 second FVC - Forced vital capacity VC - Vital capacity FEV1/VC, ratio TLC - Total lung capacity, DLCO SB - The carbon monoxide diffusion capacity (single breath method) ITGV - intrathoracic gas volume RV/TLC - Residual volume/ Total lung capacity ratio
      * validated methods of cough assessment [routine procedure]: Chung cough questionnaire and Visual analogue scale (VAS).
      * validated methods of dyspnea assessment [routine procedure]: Likert dyspnea questionnaire and modified Borg scale.

      Blood testing. In total 30 ml blood will be drawn (15 ml blood into a plain microtube without anticoagulant and 15ml blood into anticoagulation microtube). Detailed description below:

      NT-proBNP, laboratory tests performed during diagnostic process of rheumatologic diseases and potential IPAF markers [routine procedure]. 15 ml venous blood will be drawn and divided into 2 microtubes (10 ml and 5 ml) without anticoagulant 10 ml microtube will be expedited to a local laboratory in order to measure plasma levels of NT-proBNP and the following autoantibodies' titer:
      * rheumatoid factor (RF),
      * Anti-Citrullinated Protein Antibodies (ACPA; anti-CCP),
      * Antinuclear Antibodies (ANA) (ANA 1 test performed as screening); in case of ANA presence and further staining pattern identification (e.g. homogenous, speckled, peripheral, nucleolar, centromere), further tests will be performed (ANA 2 and ANA 3):

        * anti-dsDNA,
        * anti-Sm,
        * anti-SS-A (Ro),
        * anti-SS-B (La),
        * anti-Scl-70,
        * anti-RNP,
        * anti-Jo-1 and anti-PL-7, anti-PL12,
        * anti-Mi-2,
        * anti-PM-Scl,
        * anti-MDA5. From the second 5 ml microtube, after clot has formed, ca 2,5ml serum will be drawn away with a pipette; serum will be later divided into 5 Eppendorf type microtubes (0,5 ml each). These microtubes should be labeled according to the following: first letter of the patient's name- first letter of the patient's surname/ gender F or M/date of birth DD-MM-YY/date of sample collection DD-MM-YY, e.g. AL/K/12.05.45/01.02.18. The samples will be stored in -70 °C. The samples will be collected by a courier and transported to the clinical center responsible for this part of the study. This sample will be used to test for potential IPAF markers, e.g. chemokine C-C motif ligand 18 (CXCL18), Surfactant Protein A- (SP-A), Surfactant Protein D (SP-D), Krebs von den Lungen-6 protein (KL-6) and chitotrisidase 1 (CHIT1) [non-routine procedure].

      Blood sample collection [procedure not routinely performed during clinical care]. 15 ml of whole venous blood will be drawn and then divided into 10 Eppendorf tubes 1, 5 ml each. The tubes will be labeled as described above. The specimens will be stored in -70 °C. The samples will be transported to the clinical center responsible for this part of the study.

      Optionally, additional tests (testing for proteomic and metabolomic biomarkers) will be performed in samples of biological material collected beforehand (BALF, serum, urine [non-routine procedure].

      o Bronchofiberoscopy with bronchalveolar lavage (BF + BAL), performing biopsy of the bronchi mucosa: BF + BAL [routine procedure]: before starting BF, regional anesthesia and sedation with use of lidocaine and midazolam will be performed, according to anesthesia protocols applied in respective endoscopy units. Intravenous cannula will be inserted prior to BF. During endoscopy, the patient will be monitored according to safety protocols applied in respective endoscopy units.

      Bronchoalveolar lavage will be performed in the bronchus from the middle robe of right lung or the lingula of left lung (B4, B5). Localization will be chosen based on HRCT results and will be recorded in patient's medical history. Sterile solution of 0, 9% NaCl will be instilled. 200 ml fluid will be applied with a syringe in portions of 25 ml or 50 ml. It is recommended that minimum 60 % of the lavage fluid is retrieved.

      Bronchoalveolar lavage fluid (BALF) testing. Preparation of microscopic slides, analysis of the cellular components of the specimen (kind of the most abundant cells retrieved, the cells' durability) will be performed according to a standard laboratory procedure (guidelines of the Polish Respiratory Society). Total cell count along with cells' durability will be measured in a sample taken from the filtrate or material after the first spin. Cytospin (routinely 10 min of 1200-2000 rpm) will be used to prepare the material. May-Grunewald-Giemsa stain will be used to prepare the microscopic slides.

      BALF samples will be secured and stored in order to test for potential IPAF markers. 15 ml BALF will be divided into Eppendorf 1,5 ml microtubes and then stored in - 70 C. Samples will be checked for concentration of S1009A protein, chemokine (C-C motif) ligand 2 and chitotrisidase 1 (CHIT 1).

      Specimens of bronchial mucosa taken during BF [procedure not routinely performed during clinical care]. 5 mucosa specimens will be taken from the initial segment of the middle lobe bronchus, placed into Eppendorf microtubes and stored in -80 C. Specimen will be sent for histopathological assessment.
      * 6 minute walking test - (6MWT) performed according to a protocol applied in respective clinical centers [routine procedure]. The following data should be recorded:

        • Whether the patient completed the test. If 6MWT was interrupted, the reason should be recorded (e.g. dyspnea, high blood pressure, cardiac arrhythmia, intermittent claudication, other)

        • Distance in meters
        * Pulse oximetry measured before and directly after the test
        * Dyspnea measurement - Borg scale
      * High resolution computed tomography (HRCT) [routine procedure]. Current tomography, performed according to protocol applied in respective clinical centers or CT 6 months prior to the study will be eligible. Test results (saved on CD) and radiological description will be used. CD will be labeled in a way described above. OsiriX Lite software will be used to assess the scans. The following densitometric values will be measured: mean lung attenuation (MLA), kurtosis, skewness, and standard deviation of lung radiodensity (SD I.R). Data analysis will be performed with Statistica software. Data will be presented as median and interquartile ranges (IQR). Quantitative data will be analyzed with Kruskal-Willis' and Dunn's post hoc tests
      * Pulse oximetry (SpO2) [routine procedure]. If SpO2 is measured to be < 92% or if there are indications for oxygen therapy, arterial blood gas will be performed.
      * Transthoracic echocardiography (TTE) [routine procedure] with detailed right heart assessment:

      Pulmonary artery diameter Acceleration time (Act) and pulmonary regurgitation Tricuspid annulus systolic velocity Tricuspid regurgitation velocity. Tricuspid annular plate systolic excursion, (TAPSE) Basal right ventricle (RV) diameter, mid RV diameter and base-apex dimension Right ventricle inflow tract dimension Right ventricle outflow tract dimension Right ventricle diameter measured at the level of pulmonary valve Right atrial volume Superior vena cava dimension Inferior vena cava dimension Right ventricular wall thickness (RVWT) o Rheumatology consultation of every patient in IPAF and autoimmune disorder groups [procedure routinely performed during clinical care].

      Qualification for visit 2-5 - only patients qualified to phase 2 of the study

      Visit 2:

      • 6 +/- 3 months from visit 1:
      * Visit 1-5 questionnaire [non-routine procedure]
      * Lung function tests [routine procedure]
      * 6MWT [routine procedure]
      * Pulse oximetry [routine procedure]

      Visit 3:

      • 12 +/- 3 months from visit 1:
      * Visit 1-5 questionnaire [non-routine procedure]
      * Lung function tests [routine procedure]
      * 6MWT [routine procedure]
      * HRCT [routine procedure]
      * Blood testing (basic laboratory tests [routine procedure], screening for autoantibodies and cytokine concentration [non-routine procedure]
      * BF + BAL [optionally; routine procedure]
      * Arterialized capillary blood gas [routine procedure]
      * TTE with detailed right heart assessment [routine procedure]
      * Rheumatology consultation [routine procedure]

      Visit 4:

      • 24 +/- 3 months from visit 1:
      * Visit 1-5 questionnaire [non-routine procedure]
      * Lung function tests [routine procedure]
      * 6MWT [routine procedure]
      * HRCT [routine procedure]
      * Blood testing (basic laboratory tests [routine procedure], screening for autoantibodies and cytokine concentration [non-routine procedure]
      * BF + BAL (optionally; routine procedure]
      * Arterialized capillary blood gas [routine procedure]

      Visit 5

      • 60 +/- 3 months from visit 1

      o Visit 1-5 questionnaire [non-routine procedure]

      o Lung function tests [routine procedure]

      o 6MWT [routine procedure]
      * HRCT [routine procedure]
      * Blood testing (basic laboratory tests [routine procedure], screening for autoantibodies and cytokine concentration [non-routine procedure]
      * BF + BAL (optionally; routine procedure)
      * Arterialized capillary blood gas testing [routine procedure]
      * TTE with detailed right heart assessment [routine procedure]
      * Rheumatology consultation [routine procedure]
      * Optionally, in case of clinical and/or radiological progression, worsening of lung function tests' results, criobiopsy. may be repeated after obtaining informed patient consent.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent to participate in the study
* diagnosis of one of interstitial lung diseases/autoimmune diseases as described below

Exclusion Criteria:

* age < 18 years
* withdrawal od consent
* pregnancy
* lactation
* infectious disease 4 weeks prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from patients hospitalized in pneumonology wards in clinical centers participating in the study. They will be divided into 3 subgroups:
  Study group - IPAF. 2. Control groups:
  1. Connective tissue disease associated interstitial lung disease (CTD-ILD) patients:
  2. Idiopathic interstitial pneumonia group
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2019-03-18 (Estimated); Primary Completion 2020-02-18 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of IPAF diagnostic markers | 10.2019-10.2020
  It is still unclear whether there are diagnostic markers specific for IPAF or whether there is a significant difference in concentration of fibrosis biomarkers in IPAF, CTD-ILD and ILD groups. Both blood and BAL biomarkers will be taken under consideration, they include chemokine C-C motif ligand 18 (CXCL18), Surfactant Protein A- (SP-A), Surfactant Protein D (SP-D), Krebs von den Lungen-6 protein (KL-6) and chitotrisidase 1 (CHIT1).

CONTACTS AND LOCATIONS:
Overall Officials: Szymon Skoczynski, MD, PhD, Study Chair — Slaski Uniwersytet Medyczny
Locations (7):
- Universita' degli Studi di Messina, Messina, Province Of Messina, Italy
- Poland (6):
  - Katedra i Klinika Pulmonologii, Alergologii i Onkologii Pulmonologicznej Uniwersytetu Medycznego im. K. Marcinkowskiego w Poznaniu, Poznan, Greater Poland Voivodeship
  - II Katedra Chorob Wewnetrznych Uniwersytetu Jagiellonskiego Collegium Medicum im. prof. A. Szczeklika Szpitala Uniwersyteckiego, Krakow, Lesser Poland Voivodeship
  - Katedra i Klinika Pneumonologii, Onkologii i Alergologii Uniwersytetu Medycznego w Lublinie, Lublin, Lublin Voivodeship
  - Klinika Alergologii Gdanskiego Uniwersytetu Medycznego, Gdansk, Pomeranian Voivodeship
  - Katedra i Klinika Pneumonologii Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice, Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 im. prof. St. Szyszko Sląskiego Uniwersytetu Medycznego w Katowicach, Zabrze, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rzepka-Wrona P, Skoczynski S, Barczyk A. Are There Differences in Inflammatory and Fibrotic Pathways between IPAF, CTD-ILDs, and IIPs? A Single-Center Pilot Study. Int J Mol Sci. 2022 Dec 2;23(23):15205. doi: 10.3390/ijms232315205. PMID 36499525